CLINICAL TRIAL: NCT02382601
Title: Longitudinal Study of Intra-Uterine Growth Restriction (IUGR)
Brief Title: Longitudinal Study of Intra-Uterine Growth Restriction
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Perelman Family Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 14-1360
Record Dates: First submitted 2015-03-02; First posted 2015-03-09 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: IUGR; Pregnancy
Keywords: Pregnancy; IUGR; Small for gestational age
MeSH Terms: interventions — High-Energy Shock Waves; Blood Specimen Collection; PEAPOD protein, Arabidopsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal peripheral blood and umbilical cord blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Small for Gestational Age Pregancies (controls): Small for gestational age (SGA) pregnancies that do not develop IUGR will be considered controls. Each subject will have an ultrasound, MRI, maternal blood and cord blood collection, placental analysis, neurological function assessments (infant), and body fat measurements (infant).
  Interventions: Radiation: Ultrasound; Radiation: MRI; Procedure: Blood collection; Behavioral: Neurological Function Assessment; Procedure: Placental Analysis; Procedure: Measurement of body fat; Radiation: Pediatric heart ultrasound
- IUGR Pregnancies (cases): Small for gestational age (SGA) pregnancies that do develop IUGR will be considered cases. Each subject will have an ultrasound, MRI, maternal blood and cord blood collection, placental analysis, neurological function assessments (infant), and body fat measurements (infant).
  Interventions: Radiation: Ultrasound; Radiation: MRI; Procedure: Blood collection; Behavioral: Neurological Function Assessment; Procedure: Placental Analysis; Procedure: Measurement of body fat; Radiation: Pediatric heart ultrasound

INTERVENTIONS:
Radiation: Ultrasound — With 3-D and 4-D high-resolution color Doppler methods it is possible to map out the placental circulation, fetal circulation, fetal brain, and fetal cardiac function. Investigators will collect these data points prenatally.
Radiation: MRI — Similar to the Ultrasound data, investigators will collect MRI images of the fetal brain and the placenta. MRI will allow investigators to collect more detailed images of both the fetal brain and placenta, and investigators will be utilizing this technique both prenatally and postnatally.
Procedure: Blood collection — The maternal and cord blood will be collected for the processing of plasma and serum. There may be early biomarkers of IUGR in the maternal circulation that investigators can use to better determine the appropriate strategy for clinical management of care. Collection and subsequent analysis of molecular markers in the umbilical cord blood will be used to further confirm physiological dysfunction as detected by ultrasound and MRI techniques.
Behavioral: Neurological Function Assessment — Neurological development tests including a Bayley exam, Mullen exam, Developmental Profile-3, Child Behavior Checklist, and Pediatric Stroke Outcome Measure (PSOM) will be performed.
Procedure: Placental Analysis — Placentas will undergo pathological evaluation for placental function.
Procedure: Measurement of body fat — The baby's body fat will be measured in a special incubator called a PEAPOD or BODPOD when an infant.
  Other Names: Peapod; Bodpod
Radiation: Pediatric heart ultrasound — Children will have ultrasounds of their hearts during follow-up visits.

SUMMARY:
The investigation will employ a longitudinal approach in which every fetus diagnosed to be SGA (Small for Gestational Age ) will be studied at frequent intervals with sophisticated imaging techniques to assess subtle physiologic changes in the brain, heart, and placenta over time. These findings will be correlated with neurological and cardiovascular function in the newborn and early childhood. This research initiative should yield diagnostic and therapeutic templates that will improve the quality of life of IUGR babies in addition to providing important information that will better inform current diagnostic practices.

DETAILED DESCRIPTION:
The overarching objective is to serially assess changes in the fetal circulation, heart, and brain with sophisticated ultrasound, MRI (Magnetic Resonance Imaging), and body composition techniques that will provide clues as to how growth restricted babies will tolerate life outside the uterus. Employing a longitudinal study will allow the investigators to correlate perinatal and postnatal outcomes more comprehensively than previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed SGA by an ultrasound estimated fetal weight (EFW) of less than the 10th percentile or a fetal abdominal circumference of less than the 5th percentile will be included in the study at the time of their first examination.

Exclusion Criteria:

* Patients < 18 years of age, and chromosomal anomalies as identified by regular aneuploidy screening.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: University of Colorado School of Medicine is a referral center for women carrying fetuses with IUGR. Care providers routinely evaluate more than 300 patients per year at our outreach sites alone whose fetuses have estimated fetal weights below the 10th percentile. Of these, the investigators will initially enroll 200 patients per year between 24 and 36 weeks over a two-year period.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Characterize the sequence of neurological and cardiovascular events defining early and late IUGR pathogenesis, respectively | Every two weeks from the time of IUGR diagnosis or first visit
  Using ultrasound and MRI to identify changes in the fetal vasculature, and fetal brain as early and late IUGR progress.

SECONDARY OUTCOMES:
Correlate in utero adaptations in early and late IUGR, to infant and early childhood neurodevelopment | Baseline (Day 0), 40-44 weeks gestational age (post-birth), 6 months, 1-7 years
  Assess neurodevelopment with a series of tests (PSOM, Bayleys III, Mullen's Scale of Early Learning, Developmental Profile-3, Child Behavior Checklist) and correlate neurological in utero findings to neurodevelopment outcomes after birth.
Correlate in utero adaptations in early and late IUGR, to infant and early childhood cardiovascular outcomes | Baseline (Day 0), 40-44 weeks gestational age (post-birth), 6 months, 1-7 years
  Assess cardiovascular health via heart ultrasound after birth
Correlate in utero adaptations in early and late IUGR, to infant and early childhood metabolic outcomes | Baseline (Day 0), 40-44 weeks gestational age (post-birth), 6 months, 1-7 years
  Correlate IUGR severity to metabolic outcomes as assessed by body composition (pea pod and bod pod with a pediatric attachment), anthropometrics, and a diet questionnaire after birth.
Compare early IUGR, late IUGR and SGA infant and early childhood outcomes | Baseline (Day 0), 40-44 weeks gestational age (post-birth), 6 months, 1-7 years
  Using the tests describe above compare the outcomes of each group after birth.

CONTACTS AND LOCATIONS:
Overall Officials: John Hobbins, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Background] Barker ED, McAuliffe FM, Alderdice F, Unterscheider J, Daly S, Geary MP, Kennelly MM, O'Donoghue K, Hunter A, Morrison JJ, Burke G, Dicker P, Tully EC, Malone FD. The role of growth trajectories in classifying fetal growth restriction. Obstet Gynecol. 2013 Aug;122(2 Pt 1):248-254. doi: 10.1097/AOG.0b013e31829ca9a7. PMID 23969791
- [Background] Mongelli M, Gardosi J. Reduction of false-positive diagnosis of fetal growth restriction by application of customized fetal growth standards. Obstet Gynecol. 1996 Nov;88(5):844-8. doi: 10.1016/0029-7844(96)00285-2. PMID 8885925
- [Background] Cruz-Martinez R, Figueras F, Hernandez-Andrade E, Puerto B, Gratacos E. Longitudinal brain perfusion changes in near-term small-for-gestational-age fetuses as measured by spectral Doppler indices or by fractional moving blood volume. Am J Obstet Gynecol. 2010 Jul;203(1):42.e1-6. doi: 10.1016/j.ajog.2010.02.049. Epub 2010 May 1. PMID 20435282
- [Background] Hecher K, Bilardo CM, Stigter RH, Ville Y, Hackeloer BJ, Kok HJ, Senat MV, Visser GH. Monitoring of fetuses with intrauterine growth restriction: a longitudinal study. Ultrasound Obstet Gynecol. 2001 Dec;18(6):564-70. doi: 10.1046/j.0960-7692.2001.00590.x. PMID 11844190
- [Background] Ferrazzi E, Bozzo M, Rigano S, Bellotti M, Morabito A, Pardi G, Battaglia FC, Galan HL. Temporal sequence of abnormal Doppler changes in the peripheral and central circulatory systems of the severely growth-restricted fetus. Ultrasound Obstet Gynecol. 2002 Feb;19(2):140-6. doi: 10.1046/j.0960-7692.2002.00627.x. PMID 11876805
- [Background] Turan OM, Turan S, Berg C, Gembruch U, Nicolaides KH, Harman CR, Baschat AA. Duration of persistent abnormal ductus venosus flow and its impact on perinatal outcome in fetal growth restriction. Ultrasound Obstet Gynecol. 2011 Sep;38(3):295-302. doi: 10.1002/uog.9011. PMID 21465604
- [Background] Acharya G. Measurement of atrioventricular annular plane displacement has been revived: will it prove to be useful in assessing fetal cardiac function? Ultrasound Obstet Gynecol. 2013 Aug;42(2):125-9. doi: 10.1002/uog.12542. No abstract available. PMID 23775904
- [Background] Kiserud T. Re: umbilical vein flow and perinatal outcome in term small-for-gestational-age fetuses. M. Parra-Saavedra, F. Crovetto, S. Triunfo, S. Savchev, G. Parra, M. Sanz, E. Gratacos and F. Figueras. Ultrasound Obstet Gynecol 2013; 42: 189-195. Ultrasound Obstet Gynecol. 2013 Aug;42(2):130. doi: 10.1002/uog.12553. No abstract available. PMID 23893598
- [Background] Odibo AO, Zhong Y, Longtine M, Tuuli M, Odibo L, Cahill AG, Macones GA, Nelson DM. First-trimester serum analytes, biophysical tests and the association with pathological morphometry in the placenta of pregnancies with preeclampsia and fetal growth restriction. Placenta. 2011 Apr;32(4):333-8. doi: 10.1016/j.placenta.2011.01.016. Epub 2011 Feb 13. PMID 21324404
- [Background] Hafner E, Metzenbauer M, Stumpflen I, Waldhor T. Measurement of placental bed vascularization in the first trimester, using 3D-power-Doppler, for the detection of pregnancies at-risk for fetal and maternal complications. Placenta. 2013 Oct;34(10):892-8. doi: 10.1016/j.placenta.2013.06.303. Epub 2013 Jul 24. PMID 23890468
- [Background] Egana-Ugrinovic G, Sanz-Cortes M, Figueras F, Bargallo N, Gratacos E. Differences in cortical development assessed by fetal MRI in late-onset intrauterine growth restriction. Am J Obstet Gynecol. 2013 Aug;209(2):126.e1-8. doi: 10.1016/j.ajog.2013.04.008. Epub 2013 Apr 9. PMID 23583839
- [Background] Figueras F, Cruz-Martinez R, Sanz-Cortes M, Arranz A, Illa M, Botet F, Costas-Moragas C, Gratacos E. Neurobehavioral outcomes in preterm, growth-restricted infants with and without prenatal advanced signs of brain-sparing. Ultrasound Obstet Gynecol. 2011 Sep;38(3):288-94. doi: 10.1002/uog.9041. Epub 2011 Aug 10. PMID 21557369
- [Background] Eixarch E, Meler E, Iraola A, Illa M, Crispi F, Hernandez-Andrade E, Gratacos E, Figueras F. Neurodevelopmental outcome in 2-year-old infants who were small-for-gestational age term fetuses with cerebral blood flow redistribution. Ultrasound Obstet Gynecol. 2008 Dec;32(7):894-9. doi: 10.1002/uog.6249. PMID 19035538
- [Background] Fowlkes JB, Holland CK. Mechanical bioeffects from diagnostic ultrasound: AIUM consensus statements. American Institute of Ultrasound in Medicine. J Ultrasound Med. 2000 Feb;19(2):69-72. doi: 10.7863/jum.2000.19.2.69. No abstract available. PMID 10680613
- [Background] Torloni MR, Vedmedovska N, Merialdi M, Betran AP, Allen T, Gonzalez R, Platt LD; ISUOG-WHO Fetal Growth Study Group. Safety of ultrasonography in pregnancy: WHO systematic review of the literature and meta-analysis. Ultrasound Obstet Gynecol. 2009 May;33(5):599-608. doi: 10.1002/uog.6328. PMID 19291813
- [Background] Ang ES Jr, Gluncic V, Duque A, Schafer ME, Rakic P. Prenatal exposure to ultrasound waves impacts neuronal migration in mice. Proc Natl Acad Sci U S A. 2006 Aug 22;103(34):12903-10. doi: 10.1073/pnas.0605294103. Epub 2006 Aug 10. PMID 16901978
- [Background] Salvesen KA, Eik-Nes SH. Ultrasound during pregnancy and subsequent childhood non-right handedness: a meta-analysis. Ultrasound Obstet Gynecol. 1999 Apr;13(4):241-6. doi: 10.1046/j.1469-0705.1999.13040241.x. PMID 10341401
- [Background] Newnham JP, Doherty DA, Kendall GE, Zubrick SR, Landau LL, Stanley FJ. Effects of repeated prenatal ultrasound examinations on childhood outcome up to 8 years of age: follow-up of a randomised controlled trial. Lancet. 2004 Dec 4-10;364(9450):2038-44. doi: 10.1016/S0140-6736(04)17516-8. PMID 15582061
- [Background] Schwartz JL, Crooks LE. NMR imaging produces no observable mutations or cytotoxicity in mammalian cells. AJR Am J Roentgenol. 1982 Sep;139(3):583-5. doi: 10.2214/ajr.139.3.583. No abstract available. PMID 6981326
- [Background] Thomas A, Morris PG. The effects of NMR exposure on living organisms. I. A microbial assay. Br J Radiol. 1981 Jul;54(643):615-21. doi: 10.1259/0007-1285-54-643-615. PMID 6455175
- [Background] Baker PN, Johnson IR, Harvey PR, Gowland PA, Mansfield P. A three-year follow-up of children imaged in utero with echo-planar magnetic resonance. Am J Obstet Gynecol. 1994 Jan;170(1 Pt 1):32-3. doi: 10.1016/s0002-9378(94)70379-5. PMID 8296840
- [Background] Simon EM, Goldstein RB, Coakley FV, Filly RA, Broderick KC, Musci TJ, Barkovich AJ. Fast MR imaging of fetal CNS anomalies in utero. AJNR Am J Neuroradiol. 2000 Oct;21(9):1688-98. PMID 11039352
- [Background] Runge VM. Safety of approved MR contrast media for intravenous injection. J Magn Reson Imaging. 2000 Aug;12(2):205-13. doi: 10.1002/1522-2586(200008)12:23.0.co;2-p. PMID 10931582
- [Background] Victoria T, Jaramillo D, Roberts TP, Zarnow D, Johnson AM, Delgado J, Rubesova E, Vossough A. Fetal magnetic resonance imaging: jumping from 1.5 to 3 tesla (preliminary experience). Pediatr Radiol. 2014 Apr;44(4):376-86; quiz 373-5. doi: 10.1007/s00247-013-2857-0. Epub 2014 Mar 27. PMID 24671739
- [Background] Savchev S, Figueras F, Cruz-Martinez R, Illa M, Botet F, Gratacos E. Estimated weight centile as a predictor of perinatal outcome in small-for-gestational-age pregnancies with normal fetal and maternal Doppler indices. Ultrasound Obstet Gynecol. 2012 Mar;39(3):299-303. doi: 10.1002/uog.10150. Epub 2012 Feb 7. PMID 22102177
- [Background] Chawengsettakul S, Russameecharoen K, Wanitpongpan P. Fetal cardiac function measured by myocardial performance index of small-for-gestational age fetuses. J Obstet Gynaecol Res. 2015 Feb;41(2):222-8. doi: 10.1111/jog.12508. Epub 2014 Aug 27. PMID 25158601
- [Background] Mailath-Pokorny M, Worda K, Schmid M, Polterauer S, Bettelheim D. Isolated single umbilical artery: evaluating the risk of adverse pregnancy outcome. Eur J Obstet Gynecol Reprod Biol. 2015 Jan;184:80-3. doi: 10.1016/j.ejogrb.2014.11.007. Epub 2014 Nov 20. PMID 25463640